CLINICAL TRIAL: NCT02329132
Title: Change Oxygen Consumption Following Intravitreal Treatment of Lucentis (Ranibizumab) in Eyes With Diabetic Macular Edema
Status: Completed | Type: Observational
Sponsor: Kagawa University (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Akitaka Tsujikawa, Professor and Chairman, Kagawa University
Other Study IDs: H26-000
Record Dates: First submitted 2014-12-26; First posted 2014-12-31 (Estimated); Last update posted 2018-03-08 (Actual); Status verified 2018-03

CONDITIONS: Diabetic Macular Edema
Keywords: diabetic macular edema; VEGF; ranibizumab; oxygen consumption
MeSH Terms: interventions — Ranibizumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Aqueous humor is obtained at the initial injection of Lucentis.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ranibizumab — Each eye will be treated with three initial monthly injections of intravitreal ranibizumab 0.5 mg (Lucentis), followed by retreatment as needed, guided by monthly clinical examinations including biomicroscopy, VA measurement, and optical coherence tomography (OCT) examination.
  Other Names: Lucentis

SUMMARY:
Recent reports suggest that anti-VEGF agents (ranibizumab) may suppress the progression of retinal nonperfusion area. This protective effect would cause the increase of the oxygen consumption in the diabetic retina. We expect that the current study using the retinal oximetry would show the protective effects of ranibizumab on the hypoxia in the diabetic retina. This study is designed to analyze the effects of ranibizumab (Lucentis) to the retinal oxygen saturation or consumption in eyes with diabetic macular edema.

DETAILED DESCRIPTION:
Diabetic retinopathy is characterized by the retinal non-perfusion areas (the retinal hypoxia), leading to the upregulation of vascular endothelial growth factors (VEGF). Subsequently, VEGF causes increased vascular leakage, retinal vasodilation, and the development of macular edema. Based on these mechanisms, the oxygen saturation in the retinal vessels or retinal oxygen consumption would reflect the degree of underlying retinal hypoxia. Injections of anti-VEGF agents (ranibizumab) reduce the macular edema and may suppress the progression of retinal nonperfusion area. However, so far, limited information is available on the effects of anti-VEGF agents (ranibizumab) to the retinal hypoxic conditions. In addition, baseline conditions of the oxygen saturation in the retinal vessels may provide us the predictive information on the treatment efficacy of anti-VEGF agents (ranibizumab) to the diabetic macular edema.

Recent reports suggest that anti-VEGF agents (ranibizumab) may suppress the progression of retinal nonperfusion area. This protective effect would cause the increase of the oxygen consumption in the diabetic retina. We expect that the current study using the retinal oximetry would show the protective effects of ranibizumab on the hypoxia in the diabetic retina.

In addition, previous studies showed an increased VEGF level in the aqueous humor or the vitreous, depending on the progression of the diabetic retinopathy. The level of VEGF in the aqueous humor would reflect the retinal hypoxia and may be of use for the prediction of the visual prognosis. This study is designed to analyze the effects of ranibizumab (Lucentis) to the retinal oxygen saturation or consumption in eyes with diabetic macular edema.

Each eye will be treated with three initial monthly injections of intravitreal ranibizumab 0.5 mg (Lucentis), followed by retreatment as needed, guided by monthly clinical examinations including biomicroscopy, VA measurement, and optical coherence tomography (OCT) examination. The principal criteria for retreatment are the reduction of VA, foveal and extrafoveal macular edema or serous retinal detachment on OCT.

At each visit, both eyes are scheduled to be examined with VA measurement, OCT examination, oxygen saturation measurement. Just before the first injection of ranibizumab, aqueous humor will be extracted with a pipet.

Retinal oximetry will be performed with Oxymap (Oxymap ehf, Reykjavik, Iceland). Briefly, the device simultaneously acquires digital images at two wavelengths and automatically tracks retinal vessels on both images. Retinal vessel oxygen saturation is estimated by spectrophotometric analysis of light reflected from retinal vessels and from the immediately surrounding retina. Oxygen saturation measurements are made on major temporal arteries and veins. Briefly, the first and second degree vessels are used, with the addition of third degree vessels in images where peripapillary haemorrhage prevented analysis close to the optic disc. Vessel segments chosen for analysis are used consistently for consecutive measurements in the same retina.

ELIGIBILITY:
Inclusion Criteria:

1. Diabetic macular edema involving the foveal center
2. Male or female of aged 18 years or older
3. Decrease of visual acuity (VA) due to macular edema
4. Signed informed consent form

Exclusion Criteria:

1. Previous treatment with anti-VEGF drugs or corticosteroid or grid laser photocoagulation
2. Ocular disorders in the study eye that may confound interpretation of study results
3. History of vitrectomy surgery, or other surgical intervention other than the cataract surgery
4. The pregnant or lactating woman

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Diabetic macular edema involving the foveal center, who are planned to be treated with intravitreal injections of ranibizumab.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2015-11; Primary Completion 2018-01-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
The change of retinal oxygen saturation and consumption from baseline at 6 months | At 6 months after ranibizumab (Lucentis) treatment.
  Retinal oximetry will be performed with Oxymap (Oxymap ehf, Reykjavik, Iceland). Briefly, the device simultaneously acquires digital images at two wavelengths and automatically tracks retinal vessels on both images. Retinal vessel oxygen saturation is estimated by spectrophotometric analysis of light reflected from retinal vessels and from the immediately surrounding retina. Oxygen saturation measurements are made on major temporal arteries and veins. Briefly, the first and second degree vessels are used, with the addition of third degree vessels in images where peripapillary haemorrhage prevented analysis close to the optic disc. Vessel segments chosen for analysis are used consistently for consecutive measurements in the same retina. Oxygen saturation measurements will be measured at each visit for 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: AKITAKA TSUJIKAWA, MD, Principal Investigator — Kagawa Univerisity Faculty of Medicine
Locations (1):
- Kagawa University Faculty of Medicine, Hiragi, Kagawa-ken, Japan